CLINICAL TRIAL: NCT06153537
Title: A Multi-centre, Prospective, Non-interventional, Single-arm Study Investigating Glycaemic Control Associated With the Use of Dose Check App and Insulin Degludec in Patients With Type 2 Diabetes Mellitus in Saudi Arabia Under Real-world Setting
Brief Title: A Research Study in Saudi Arabia to Understand How the Dose Check App Used With Tresiba Treatment Helps to Control Blood Sugar Level
Acronym: DEAL-2
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1250-7588; U1111-1288-8138 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-11-23; First posted 2023-12-01 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Insulin degludec + dose check: Participants will be treated with commercially available insulin degludec used with Dose Check app according to local label and routine clinical practice at the discretion of the treating physician.
  Interventions: Drug: Insulin degludec

INTERVENTIONS:
Drug: Insulin degludec — Participants will be treated with commercially available insulin degludec used with Dose Check app according to local label and routine clinical practice at the discretion of the treating physician.
  Other Names: Tresiba

SUMMARY:
This study looks at how a mobile based app called 'Dose Check' used along with Tresiba helps to control blood sugar level in participants with type 2 diabetes mellitus. Participants will get Tresiba as prescribed by the study doctor or participants will continue already prescribed treatment with Tresiba. Participants will also be prescribed to use Dose Check app by the study doctor and will be asked to install the Dose Check app in their mobile phone, which will support participants with the correct dose of Tresiba. This study will last for about 6 to 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Male or female, age above or equal to 21 years at the time of signing informed consent.
* Diagnosed with type 2 diabetes mellitus (T2DM) above or equal to 12 weeks prior to signing consent.
* The decision to initiate treatment with commercially available Dose Check app as a part of treatment along with Tresiba as per the local label, has been made by the participant and the treating physician before and independently from the decision to include the participant in this study.
* Available HbA1c value less than or equal to 12 weeks prior to the 'Informed consent and initiation of Dose Check app visit' (V1) or HbA1c measurement taken in relation with the 'Informed consent and initiation of Dose Check app visit (V1)' (V1) or planned soon after V1 (less than or equal to 7 days), if in line with local clinical practice.
* Willingness to continue using the Dose Check app on a compatible smartphone according to the intended use for the entire duration of the study.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having signed informed consent in this study.
* Women known to be pregnant or breastfeeding, or women planning to become pregnant during the conduct of the study.
* Treatment with any investigational drug or software as medical device (SaMD) within 30 days prior to enrolment into the study.
* Diagnosed with type 1 diabetes mellitus.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Hypersensitivity to the active substance or any of the excipients as specified in the Tresiba local label.
* On treatment with Tresiba for above 3 months or at dose above 20 units at Informed consent and initiation of Dose Check app visit (V1).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with T2DM and aged less than or equal to 21 years.
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to end of study visit(week 26 [-4 to +8 weeks])
  Measured in percentage point.

SECONDARY OUTCOMES:
Participants reaching individual HbA1c target set by physician | end of study visit (week 26 [-4 to +8 weeks])
  Measured as number of participants (yes/no).
Participants reaching physician set individual fasting blood glucose (FBG) target | From baseline (week 0) to end of study visit(week 26 [-4 to +8 weeks])
  Measured as number of participants (yes/no).
Time to physician set individual FBG target from first reported FBG | From baseline (week 0) to end of study visit(week 26 [-4 to +8 weeks])
  Measured in weeks.
Participants achieving target level FBG according to clinical guidance | From baseline (week 0) to end of study visit(week 26 [-4 to +8 weeks])
  Measured as number of participants (yes/no).
Change in laboratory measured FPG | From baseline (week 0) to end of study visit(week 26 [-4 to +8 weeks])
  Measured in milligrams per deciliter (mg/dL).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (13):
- Saudi Arabia (13):
  - Dr. Sulaiman Al Habib- Al Qassim, Buraidah, Al Qassim
  - Almoosa Specialist Hospital, Ihsaa
  - Saudi airlines Medical Services, Jeddah
  - Saudi German Hospital, Jeddah
  - My clinic, Jeddah
  - Saudi German Hospital, Khamis Mushait
  - Al Mowasat Khobar, Khobar
  - Sulaiman Al Habib- Al Khobar, Khobar
  - King Fahad Hospital of the University, Khobar
  - Al Hammadi, Riyadh
  - Dr. Sulaiman Al Habib Medical Group- Olaya, Riyadh
  - King Fahd Medical City, Riyadh, KSA, Riyadh
  - Dr. Sulaiman Al Habib Medical Group- Swedi, Riyadh

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com